CLINICAL TRIAL: NCT03557619
Title: A Study to Assess the Effect of Venetoclax on the Pharmacokinetics of Ethinyl Estradiol/Levonorgestrel in Female Subjects With Hematologic Malignancies
Brief Title: A Study to Assess the Effect of Venetoclax on Ethinyl Estradiol and Levonorgestrel in Female Participants With Different Hematological Malignancies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: M16-185
Expanded Access: NCT03123029 (Available)
Record Dates: First submitted 2018-06-05; First posted 2018-06-15 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Hematologic Malignancies
Keywords: Cancer; Hematologic Malignancies, venetoclax; ethinyl estradiol; relapsed or refractory non-Hodgkin's lymphoma; non-Hodgkin's lymphoma
MeSH Terms: conditions — Hematologic Neoplasms; Neoplasms; Recurrence; Lymphoma, Non-Hodgkin | interventions — venetoclax; Ethinyl Estradiol-Norgestrel Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ethinyl estradiol/Levonorgestrel and Venetoclax (Experimental): Ethinyl estradiol/levonorgestrel is administered on Period 1 Day 1 and then again on Period 3 Day 1. Venetoclax is administered on Period 2 Day 1 and then daily thereafter.
  Interventions: Drug: Venetoclax; Drug: ethinyl estradiol/levonorgestrel

INTERVENTIONS:
Drug: Venetoclax — tablet; oral
  Other Names: ABT-199; GDC-0199; Venclexta
Drug: ethinyl estradiol/levonorgestrel — tablet; oral
  Other Names: Levora

SUMMARY:
A study to assess the effect of multiple doses of venetoclax on the pharmacokinetics of ethinyl estradiol and levonorgestrel in female participants with different hematological malignancies. Upon completion of this study, participants receiving clinical benefit in the opinion of the investigator and without any clinically significant evidence of disease progression with no access to venetoclax (not approved for the treated indication) may continue receiving venetoclax at the discretion of the investigator in a separate extension study.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have relapsed or refractory non-Hodgkin's lymphoma (NHL).
* Participant must have histologically documented diagnosis of one of the following NHL subtypes: diffuse large B-cell lymphoma (DLBCL), follicular lymphoma (FL), lymphoplasmacytic lymphoma (LPL), mantle cell lymphoma (MCL), marginal zone lymphoma (MZL), T-cell prolymphocytic lymphoma (T-PLL), Waldenström's macroglobulinemia (WM)
* Has an Eastern Cooperative Oncology Group (ECOG) performance score of less than or equal to two.
* Must have adequate bone marrow, coagulation, renal and hepatic function as described in the protocol.
* A female of non-childbearing potential as described in the protocol.

Exclusion Criteria:

* History of currently active, clinically significant cardiovascular disease.
* If the participant has had prior stem cell transplantation, it must have been more than 100 days prior to start of study drug, with no graft versus host disease, and no immunosuppression therapy.
* evidence of transformation of the lymphoma immediately prior to study entry.
* Evidence of central nervous system involvement by lymphoma.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2019-07-30 (Actual); Primary Completion 2026-03-21 (Estimated); Study Completion 2026-03-21 (Estimated)

PRIMARY OUTCOMES:
Tmax of Venetoclax | Up to approximately 59 days after initial study drug dose
  Time to maximum plasma concentration (Tmax) of Venetoclax.
Tmax of (ethinyl estradiol) EE/Levonorgestrel | Up to approximately 59 days after initial study drug dose
  Time to maximum plasma concentration (Tmax) of EE/Levonorgestrel
Cmax of Venetoclax | Up to approximately 59 days after initial study drug dose
  Maximum plasma concentration (Cmax) of Venetoclax
Cmax of EE/Levonorgestrel | Up to approximately 59 days after initial study drug dose
  Maximum plasma concentration (Cmax) of EE/Levonorgestrel
t1/2 of Venetoclax | Up to approximately 59 days after initial study drug dose
  Terminal phase elimination half-life (t1/2) of Venetoclax.
t1/2 of EE/Levonorgestrel | Up to approximately 59 days after initial study drug dose
  Terminal phase elimination half-life (t1/2) of EE/Levonorgestrel
AUCt of Venetoclax | Up to approximately 59 days after initial study drug dose
  Area under the plasma concentration-time curve (AUC) from time 0 to time of the last measurable concentration (AUCt) of Venetoclax
AUCt of EE/Levonorgestrel | Up to approximately 59 days after initial study drug dose
  Area under the plasma concentration-time curve (AUC) from time 0 to time of the last measurable concentration (AUCt) of EE/Levonorgestrel
AUCinf of EE/Levonorgestrel | Up to approximately 59 days after initial study drug dose
  AUC from time 0 extrapolated to infinite time (AUCinf) of EE/Levonorgestrel.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (4):
- United States (3):
  - Duplicate_Henry Ford Health System /ID# 209090, Detroit, Michigan
  - Dartmouth-Hitchcock Medical Center /ID# 169097, Lebanon, New Hampshire
  - Gabrail Cancer Center Research /ID# 207039, Canton, Ohio
- Peter MacCallum Cancer Centre-East Melbourne /ID# 225247, East Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related info — https://www.rxabbvie.com